CLINICAL TRIAL: NCT03319953
Title: A Randomized, Double-Blind, Placebo Controlled, Two-Period Cross-Over, Proof of Activity Study to Evaluate the Effects of TAK-041 on Motivational Anhedonia as Add-On to Antipsychotics in Subjects With Stable Schizophrenia
Brief Title: A Randomized, Double-Blind, Placebo Controlled, Two-Period Cross-Over, Proof of Activity Study to Evaluate the Effects of TAK-041 on Motivational Anhedonia as Add-On to Antipsychotics in Participants With Stable Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-041-2001; U1111-1191-6915 (Other: World Health Organisation); 2017-001084-20 (EudraCT Number: European Medicines Agency); 17/YH/0195 (Registry Identifier: NRES); 03319953 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Stable Schizophrenia
Keywords: Drug therapy
MeSH Terms: interventions — TAK-041

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics (Experimental): TAK-041 40 milligram (mg), suspension, orally on Day 1 of Treatment Period 1, followed by 35 day Wash-out Period, followed by TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 2. All participants received a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
  Interventions: Drug: TAK-041; Drug: Placebo; Drug: Second Generation Antipsychotics (SGA)
- Treatment Sequence 2: Placebo/TAK-041 40 mg + Antipsychotics (Experimental): TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 1, followed by 35 days Wash-out Period, followed by TAK-041 40 mg, suspension, orally on Day 1 of Treatment Period 2. All participants received a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
  Interventions: Drug: TAK-041; Drug: Placebo; Drug: Second Generation Antipsychotics (SGA)
- Treatment Sequence 3: TAK-041 160 mg/Placebo + Antipsychotics (Experimental): TAK-041 160 mg, suspension, orally on Day 1 of Treatment Period 1, followed by 35 days Wash-out Period, followed by TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 2. All participants received stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
  Interventions: Drug: TAK-041; Drug: Placebo; Drug: Second Generation Antipsychotics (SGA)
- Treatment Sequence 4: Placebo/TAK-041 160 mg + Antipsychotics (Experimental): TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 1, followed by 35 days Wash-out Period, followed by TAK-041 160 mg, suspension, orally on Day 1 of Treatment Period 2. All participants received stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
  Interventions: Drug: TAK-041; Drug: Placebo; Drug: Second Generation Antipsychotics (SGA)

INTERVENTIONS:
Drug: TAK-041 — TAK-041 suspension
Drug: Placebo — TAK-041 placebo-matching suspension
Drug: Second Generation Antipsychotics (SGA) — Second generation antipsychotics included risperidone, paliperidone, iloperidone, quetiapine, olanzapine, ziprasidone, asenapine and lurasidone.

SUMMARY:
The purpose of the study is to determine whether motivation/reward deficits observed in schizophrenia are attenuated and whether cognitive impairment associated with schizophrenia is improved by add-on TAK-041 administration to antipsychotics in participants with stable schizophrenia.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-041. TAK-041 is being tested to treat people who have stable schizophrenia. This study will look whether motivation/reward deficits observed in schizophrenia are attenuated and whether cognitive impairment associated with schizophrenia is improved in people who take TAK-041 in addition to standard care.

The study will enroll approximately 32 patients. Participants will be randomly assigned (by chance, like flipping a coin) in 1:1 ratio to one of the two treatment sequences -which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need) to receive either TAK-041 40 mg or Placebo first and then will be crossed over to receive the opposite Intervention.

All participants will be asked to take oral suspension on Day 1 of each Period. There will be a wash-out Period of 35 days between the dosing days in Period 1 and 2.

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is approximately 126 to 154 days. Participants will make multiple visits to the clinic plus a final visit 77 days after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is on a stable dose of antipsychotics for at least 2 months as documented by medical history and assessed by site staff (other than those on the excluded medication list).
2. Meets schizophrenia criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) by the Mini International Neuropsychiatric Interview (MINI).
3. Have Positive and Negative Syndrome Scale (PANSS) total score less than or equal to (<=) 90 and PANSS Negative Symptom Factor Score ([NSFS]; Sum of PANSS N1, N2, N3, N4, N6, G7, and G16) greater than or equal to (>=) 15 at screening and baseline (Day -1).
4. Has stable Screening and baseline (Day-1) PANSS and NSFS total scores (less than [<] 20 percent [%] change).
5. Have had a structural brain magnetic resonance imaging (MRI) within the preceding year or during screening indicating no concerning structural brain abnormalities or other abnormalities that would interfere with interpretation of functional brain imaging results.

Exclusion Criteria:

1. Has a history of cancer (malignancy).
2. Has a positive alcohol and/ or positive drug screen at Screening or Day -1.
3. Is positive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, or human immunodeficiency virus (HIV) antibody/antigen (confirmatory testing is allowed; most sensitive test should take precedence).
4. Had major surgery, or donated or lost 1 unit of blood (approximately 500 milliliters [mL]) within 4 weeks prior to the pretrial/Screening Visit.
5. Has abnormal Screening or baseline laboratory values (>upper limit of normal [ULN] for the respective serum chemistries) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBILI), alkaline phosphatase (ALP), γ-glutamyl transferase (GGT) confirmed upon repeat testing, 5'-nucleotidase (Screening only), and/or abnormal urine osmolality, confirmed upon repeat testing.
6. Meets DSM-5 criteria for substance use disorder or history of alcohol abuse within 1 month prior to Screening Visit.
7. Has a history of claustrophobia or inability to tolerate mock scanner environment during habituation/screening session.
8. Fulfills any of the MRI contraindications on the site standard radiography screening document.
9. Has a history in the last year from the randomization visit or is currently receiving treatment with clozapine.
10. Has a current diagnosis of a significant psychiatric illness other than schizophrenia, per DSM-5 and is in an acute phase or episode.
11. Has a risk of suicide according to the investigator's clinical judgment (example, per C-SSRS positive answers on questions 4 or 5 or has made a suicide attempt within 6 months prior to screening visit).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Kings College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hawkins PCT, Schwarz AJ, Stone JM, Pepper F, Gilleen J, Gijsen S, Mazibuko N, Arkilo D, Yin W, Wu J, Khudyakov P, Behrje R, Rosen L, Posener J, Mehta MA, Laurenza A. The GPR139 agonist TAK-041 produces time-dependent alterations to cerebral blood flow and reward system function in patients with schizophrenia: a randomised placebo-controlled trial. Psychopharmacology (Berl). 2025 Aug 16. doi: 10.1007/s00213-025-06884-x. Online ahead of print. PMID 40817174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at single investigative sites in United Kingdom from 21 December 2017 to 06 November 2019.
Groups:
- Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics: TAK-041 40 milligram (mg), suspension, orally on Day 1 of Treatment Period 1, followed by 35 days wash-out Period, followed by TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 2. All participants received a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
Period: Period 1 (Day 1 to 14)
Arm/Group | Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics | Treatment Sequence 2: Placebo/TAK-041 40 mg + Antipsychotics | Treatment Sequence 3: TAK-041 160 mg/Placebo + Antipsychotics | Treatment Sequence 4: Placebo/TAK-041 160 mg + Antipsychotics
Started | 3 | 4 | 9 | 7
Completed (Completed = Participants who completed study treatment.) | 3 | 4 | 9 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (Day 15 to 49)
Arm/Group | Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics | Treatment Sequence 2: Placebo/TAK-041 40 mg + Antipsychotics | Treatment Sequence 3: TAK-041 160 mg/Placebo + Antipsychotics | Treatment Sequence 4: Placebo/TAK-041 160 mg + Antipsychotics
Started | 3 | 4 | 9 | 7
Completed | 3 | 4 | 9 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Day 49 to 154)
Arm/Group | Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics | Treatment Sequence 2: Placebo/TAK-041 40 mg + Antipsychotics | Treatment Sequence 3: TAK-041 160 mg/Placebo + Antipsychotics | Treatment Sequence 4: Placebo/TAK-041 160 mg + Antipsychotics
Started | 3 | 4 | 9 | 7
Treated (3 participants discontinued before receiving their respective treatment, per sequence, in Period 2.) | 2 | 4 | 8 | 6
Completed (Completed = Participants who completed study treatment.) | 2 | 4 | 8 | 6
Not Completed | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: TAK-041 40 mg/Placebo + Antipsychotics | Treatment Sequence 2: Placebo/TAK-041 40 mg + Antipsychotics | Treatment Sequence 3: TAK-041 160 mg/Placebo + Antipsychotics | Treatment Sequence 4: Placebo/TAK-041 160 mg + Antipsychotics | Total
Number analyzed (Participants) | 3 | 4 | 9 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (16.5) | 39.3 (16.1) | 46.8 (12.1) | 43.4 (9.6) | 43.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 6
  Male | 3 | 2 | 7 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 9 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 4 | 6 | 16
  White | 0 | 1 | 4 | 0 | 5
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Brief Assessment of Cognition in Schizophrenia (BACS) Composite Score at Second Testing After TAK-041 Administration
Description: BACS is a reliable and sensitive measure of cognitive function in schizophrenia. The BACS consists of items across six subtests: Verbal Memory, Digit Sequencing, Token Motor, Verbal Fluency, Symbol Coding, and Tower of London. The subtest scale scores were used to compute a composite BACS t-score of 50 (20) is the mean (standard deviation) of a relevant index population. Higher values indicate better performance. Bayesian normal linear model was used for analysis.
Time Frame: Baseline (Day -1) and Day 14
Population: Pharmacodynamic (PD) Analysis Set included all participants who received at least 1 dose of study drug and had at least 1 evaluable primary or exploratory PD measurement. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: t-scale
Groups:
- Placebo: TAK-041 placebo-matching, suspension, orally on Day 1 of Treatment Period 1 or 2. All participants took a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
- TAK-041 40 mg: TAK-041 40 mg, suspension, orally on Day 1 of Treatment Period 1 or 2. All participants took a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
- TAK-041 160 mg: TAK-041 160 mg, suspension, orally on Day 1 of Treatment Period 1 or 2. All participants took a stable dose of antipsychotics as per standard of care throughout the duration of the Treatment Period.
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
t-scale
  Baseline | 29.72 (12.867) | 27.35 (12.753) | 27.89 (8.214)
  Day 14: number analyzed (Participants) | 21 | 6 | 14
  Day 14 | 2.28 (6.963) | 5.35 (6.944) | 1.31 (5.618)
Statistical Analysis 1: Comparison: Placebo vs TAK-041 40 mg; Test type: Superiority; p = 0.2079, Bayesian Normal Linear Model — Bayesian method was used to calculate the posterior probability. High posterior probability of a difference between TAK-041 and placebo >2.0
Statistical Analysis 2: Comparison: Placebo vs TAK-041 160 mg; Test type: Superiority; p = 0.0633, Bayesian Normal Linear Model — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Blood-Oxygen-Level-Dependent (BOLD) Signal in the Average Ventral Striatum (VS) Region of Interest (ROI) Activation in the Monetary Incentive Delay (MID) Reward Task at First Testing After TAK-041 Administration
Description: Blood-oxygen-level-dependent imaging, or BOLD-contrast imaging, is a method used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time. The MID task is a reward anticipation paradigm that robustly engages the VS, a key area associated with coding incentive reward. Dysfunctional processing of reward information is associated with motivational impairments in schizophrenia. Motivational impairment is a key aspect of negative symptoms, and has been associated with reduced activity in the VS. Any change in BOLD signal that comes in fMRI is reported.
Time Frame: Day 1
Population: PD Analysis Set included all participants who received at least 1 dose of study drug and had at least 1 evaluable primary or exploratory PD measurement. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: BOLD signal
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 20 | 6 | 13
BOLD signal | 0.23 (0.396) | 0.23 (0.202) | 0.03 (0.458)
Statistical Analysis 1: Comparison: Placebo vs TAK-041 40 mg; Test type: Superiority; p = 0.1706, Bayesian Normal Linear Model — Bayesian method was used to calculate the posterior probability. High posterior probability of a difference between TAK-041 and placebo >0.09
Statistical Analysis 2: Comparison: Placebo vs TAK-041 160 mg; Test type: Superiority; p = 0.0373, Bayesian Normal Linear Model — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From the first dose of study drug up to 77 days after last dose of study drug (Up to Day 154)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
percentage of participants | 57.1 | 71.4 | 53.3

4. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Description: Clinical Laboratory parameters included tests for chemistry, hematology and urinalysis. Markedly abnormal values during treatment period were categorized as: alanine aminotransferase (ALT)>3.0 U/L*upper limit of normal(ULN),albumin<25 g/L*lower limit of normal(LLN), alkaline phosphatase >3.0 U/L*ULN, aspartate aminotransferase >3.0 U/L*ULN, bilirubin >34.2 umol/L*ULN, calcium <1.75 mmol/L, >2.88 mmol/L, chloride <75 mmol/L, >126 mmol/L, creatinine >177umol/L, gamma glutamyl transferase >3 U/L*ULN, glucose <2.8 mmol/L, >19.4 mmol/L, potassium<3 mmol/L, >6 mmol/L, sodium <130 mmol/L, >150 mmol/L,Urea <130 mmol/L, erythrocytes <0.8*LLN >1.2*ULN, hematocrit <0.8*LLN, >1.2*ULN, hemoglobin <0.8 g/L*LLN, >1.2 g/L*ULN, leukocytes <0.5 (10^9/L)*LLN, >1.5 (10^9/L)*ULN, platelets <75(10^9/L), >600(10^9/L).
Time Frame: From the first dose of study drug up to 77 days after last dose of study drug (Up to Day 154)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements At Least Once Post Dose
Description: Vital signs included oral body temperature measurement, supine and standing blood pressure, respiration rate, and pulse. Pulse and blood pressure were measured after 5 minutes supine and again at 1 and 3 minutes after standing. The markedly abnormal value (MAV) criteria for vital signs included systolic blood pressure < 85 mmHg, > 180 mmHg; diastolic blood pressure < 50 mmHg, > 110 mmHg; pulse < 50 beats/min, > 120 beats/min; temperature < 35.6 C > 37.7 C.
Time Frame: From the first dose of study drug up to 77 days after last dose of study drug (Up to Day 154)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug. Only categories with at least one participant are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
percentage of participants
  <35.6 C | 0 | 0 | 6.7
  >37.7 C | 4.8 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) at Least Once Post Dose
Description: The markedly abnormal value (MAV) criteria for 12-lead ECG parameters included ECG Mean Heart Rate < 50 beats/min, > 120 beats/min; PR Interval, Aggregate <= 80 msec, >= 200 msec; QRS Duration, Aggregate <= 80 msec, >= 180 msec; QTcB Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec); QTcF Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec).
Time Frame: From the first dose of study drug up to 77 days after last dose of study drug (Up to Day 154)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug. Categories with at least one participant are reported. Number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
percentage of participants
  ECG Mean Heart Rate: <50 beats per minute: number analyzed (Participants) | 19 | 5 | 15
  ECG Mean Heart Rate: <50 beats per minute | 0 | 0 | 6.7
  PR Interval: >=200 milliseconds: number analyzed (Participants) | 19 | 5 | 15
  PR Interval: >=200 milliseconds | 10.5 | 20.0 | 13.3
  QRS Duration: <=80 milliseconds: number analyzed (Participants) | 19 | 5 | 15
  QRS Duration: <=80 milliseconds | 36.8 | 20.0 | 33.3

7. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Treatment-emergent suicidal ideation (SI) or suicidal behavior (SB) compared to baseline will be measured by an increase in suicidal ideation category (1-5 on the C-SSRS) or suicidal behavior category (6-10 on the C-SSRS) during treatment from the maximum suicidal ideation/behavior category at baseline, or any suicidal ideation/behavior during treatment if there is none at baseline. C-SSRS is used to assess whether participant experienced suicidal ideation (1: wish to be dead; 2: non-specific active suicidal thoughts; 3: active suicidal ideation with any methods (not plan) without intent to act; 4: active suicidal ideation with some intent to act, without specific plan; 5: active suicidal ideation with specific plan and intent) and suicidal behavior (6: actual attempt; 7: interrupted attempt; 8: aborted attempt; 9: preparatory acts or behavior; 10: suicidal behavior).
Time Frame: Baseline (Day -1) and Days 14, 35 and 77
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug. Only categories with at least one participant are reported. Number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
Number analyzed (Participants) | 21 | 7 | 15
Participants
  SI-Wish to be Dead, Day -1 | 3 | 0 | 1
  SI-Wish to be Dead, Day 14: number analyzed (Participants) | 21 | 7 | 14
  SI-Wish to be Dead, Day 14 | 1 | 0 | 0
  SI-Wish to be Dead, Day 77: number analyzed (Participants) | 10 | 4 | 6
  SI-Wish to be Dead, Day 77 | 1 | 0 | 1
  SB-Non-suicidal Self-injurious Behaviour, Day 77: number analyzed (Participants) | 0 | 4 | 6
  SB-Non-suicidal Self-injurious Behaviour, Day 77 |  | 1 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 77 days after last dose of study drug (Up to Day 154)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | Placebo | TAK-041 40 mg | TAK-041 160 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/7 | 0/15
Other Adverse Events (participants affected / at risk) | 12/21 | 5/7 | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | TAK-041 40 mg (N=7) | TAK-041 160 mg (N=15)
Headache (Nervous system disorders) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 1
Catheter Site Pain (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Panic Attack (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Headache (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pregnancy Of Partner (Social circumstances) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03319953/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03319953/SAP_001.pdf